CLINICAL TRIAL: NCT04334421
Title: APEMESH- Preventing Perineal Complications After Abdominoperineal Resection
Status: Completed | Type: Observational
Sponsor: Elisa Mäkäräinen (Other)
Responsible Party: Sponsor-Investigator, Elisa Mäkäräinen, Principal Investigator, University of Oulu
Organization: University of Oulu (Other)
Other Study IDs: 57/2020
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Rectal Cancer; Abdominoperineal Resection; Wound Heal
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mesh group: After resection, pelvic floor is reconstructed by synthetic composite mesh (Symbotex, Medtronic) and covered with subcutaneous flap.
  Interventions: Device: Composite mesh

INTERVENTIONS:
Device: Composite mesh — Pelvic floor is reconstructed by synthetic composite mesh (Symbotex, Medtronic) to improve healing and prevent perineal herniation.

SUMMARY:
Abdominoperineal resection leaves an empty space to be filled by mesh or musculocutaneus flap. Several studies have reported over 30% morbidity with perineal wound healing after abdominoperineal resection. Preoperative radiotherapy is a strong predictor for perineal complications. Musculocutaneus flaps and use of biological mesh seem to minimize perineal morbidity. The role of omentoplasty at APR is controversial.

Previous studies on synthetic mesh repair on perineum are almost lacking.

DETAILED DESCRIPTION:
The objective of this pilot study is to assess the feasibility and the potential benefits of synthetic mesh reconstruction in perineum in case-control setting.

30 subjects will be prospectively enrolled to this study as intervention group. Controls matched with age, gender and preoperative radiotherapy are selected from retrospective data collected from Oulu University database and operated for rectal adenocarcinoma 2009-2017 with otherwise identical methods.

ELIGIBILITY:
Inclusion Criteria:

* Abdominoperineal resection and permanent colostoma

Exclusion Criteria:

* Patient with a comorbid illness of condition that would preclude the use of surgery (ASA5)
* Potentially curable resection not possible
* Patient undergoing emergency procedure
* Metastatic disease
* Pregnant or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study patients who have abdominoperineal resection
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Comprehensive Complication index | 30 days
  Comprehensive Complication index is used to evaluate outcome

SECONDARY OUTCOMES:
Surgical site infection | 30 days
  Surgical site infection classified by Clavien-Dindo score
Reoperation rate | 30 days
  Reoperations during primary stay at the hospital
Operative time | 30 days
  Operative time
Length of stay | 30 days
  Length of stay at the hospital during primary operation and recovery
Costs | 30 days
  Costs by materials used
Total perineal healing time | 30 days
  Time to point when perineum is closed and healed
Perineal sinus | 30 days
  Presence of perineal sinus at 30 days follow-up
Perineal hernia | 12 months
  Perineal hernia by CT scan at 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Mäkäräinen-Uhlbäck, M.D., Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No